CLINICAL TRIAL: NCT02760992
Title: Steady-State Bioequivalence Study of Multiple Doses of Oral Versus Intravenous Baclofen in Healthy Adult Volunteers
Brief Title: Repeated Dose IV Baclofen Safety/Bioequivalence Study
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Allaysis, LLC (Industry)
Collaborators: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CTSI - 24347
Record Dates: First submitted 2016-02-26; First posted 2016-05-04 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Intravenous Baclofen
MeSH Terms: interventions — Baclofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral Baclofen (Active Comparator): Subject will start baclofen at a 5 mg oral dose every 8 hours. Oral baclofen will be increased incrementally and self-administered over 13 days to a maximum dose of 20 mg every 8 hours. Following IV administration, subjects will be changed back to oral baclofen at a 15 mg dose self-administered every 8 hours and tapered off of baclofen over 15 days.
  Interventions: Drug: Oral Baclofen
- IV Baclofen (Experimental): Subjects will be crossed over to 16 mg intravenous baclofen infused over 120 or 150 minutes every 8 hours for 11 doses.
  Interventions: Drug: IV Baclofen

INTERVENTIONS:
Drug: IV Baclofen — Baclofen intravenous solution 2 mg/mL manufactured and provided by Allaysis, LLC
  Arms: IV Baclofen
Drug: Oral Baclofen — 10 mg tablet
  Arms: Oral Baclofen

SUMMARY:
The purpose of this study is to identify a suitable dosing regimen of IV baclofen to serve as a temporary substitute for an oral regimen.

DETAILED DESCRIPTION:
Baclofen intravenous solution 2 mg/mL will be manufactured and provided by Allaysis, LLC. Prism Clinical Research will purchase oral baclofen tablets (10 mg) from a commercial supplier. Subject will start baclofen at a 5 mg oral dose every 8 hours. Oral baclofen will be increased incrementally and self-administered over 13 days to a maximum dose of 20 mg every 8 hours. Subjects will be crossed over to 16 mg intravenous baclofen infused over 120 (n=6) or 150 (n=6) minutes every 8 hours for 11 doses. Subjects will be changed back to oral baclofen at a 15 mg dose self-administered every 8 hours and tapered off of baclofen over 15 days. Following the completion of this group of 12 subjects, the remaining 30 subjects will receive IV baclofen at the infusion duration that best meets the criteria for bioequivalence.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between the ages of 18-45. An attempt will be made to recruit an equal number of men and women into each dosing group; however a ratio of 2:4 in the initial run-in phase and 12:18, with either women or men in the majority is acceptable.
* Subjects are capable of giving informed consent.
* Females capable of bearing children should practice at least one or more of the following methods of contraception for at least one month prior to the and during the study: hormonal, intrauterine device (IUD), or barrier method in combination with a spermicide. Female subjects who are postmenopausal (no menses for greater than one year) or surgically incapable of bearing children may participate.
* Subject should be medication free, other than hormonal birth control, for 48 hours before through 24 hours after completion of study drug administration. If the need for medication is identified during this time period, it will be discussed with and approved by the PI.

Exclusion Criteria:

* Women who are pregnant.
* Women who are breastfeeding.
* Subject has a history of intolerance to IV administration of medication.
* Subject has a known hypersensitivity to baclofen.
* Subject has a significant history of cardiac, neurologic, psychiatric, oncologic, endocrine, metabolic, renal or hepatic disease
* Subject has taken or used any investigational drug or device in the 30 days prior to screening.
* Subject has taken either prescribed or over the counter medication, other than hormonal birth control within 48 hours prior to baclofen administration, unless approved by the Principal Investigator.
* Subject reveals clinically significant abnormalities on screening laboratory tests.
* Subject is a non-English speaker, such that ability to ascertain neurological status would require an interpreter.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2017-05; Primary Completion 2017-09 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Bioequivalence of IV Baclofen Relative to Oral at Steady State | 2 dosing intervals (total of 16 hours)
  Evaluate and confirm selected infusion rates of IV baclofen which best achieve bioequivalence to oral baclofen at steady state in healthy adults.

SECONDARY OUTCOMES:
Number of participants experiencing sedation due to the treatment measured by the sanford sleepiness scale | 3 months
  Over the course of the intervention (~3 months) subjects will be assessed using the Modified Sanford sleepiness scale prior to the first and second intravenous drug administration then every 30 minutes for four hours after drug administration. If this assessment shows that the subject is not at their baseline, assessments will continue every 30 minutes until the subject has returned to the baseline function.
Number of participants experiencing nystagmus due to the treatment. | 3 months
  Over the course of the intervention (~3 months) subjects will be assessed using the following rating scale and definitions of ataxia and nystagmus prior to the first and second intravenous drug administrations then every 30 minutes for four hours after drug administration. If this assessment shows that the subject is not at their baseline, assessments will continue every 30 minutes until the subject has returned to the baseline function.
  Nystagmus:
  0 = None
  1. mild - present only on extreme gaze (beyond 45 degrees lateral gaze)
  2. severe - present on neutral to 45 degrees lateral gaze
Number of participants experiencing ataxia due to the treatment measured by tandem gait | 3 months
  Over the course of the intervention (~3 months) subjects will be assessed using the following rating scale and definitions of ataxia and nystagmus prior to the first and second intravenous drug administrations then every 30 minutes for four hours after drug administration. If this assessment shows that the subject is not at their baseline, assessments will continue every 30 minutes until the subject has returned to the baseline function.
  Ataxia: For those who are ambulatory, this will be assessed by gait. Ratings will be: 0=none
  1. Mild - unsteady with tandem gait testing, but able to perform without assistance
  2. Severe - unable to perform gait testing without assistance. For non-ambulatory subjects, ataxia will be assessed by finger to nose and finger pursuit maneuvers.
Peak Plasma Concentration (Cmax) | 3 months
  Cmax will be determined on visual observation.
Area Under the Curve (AUC) | 3 months
  Pharmacokinetic analysis will be performed with WinNonLin (Pharsight), a pharmacokinetic data analysis package, and will include calculation of the area under the concentration-time curve (AUC).

IPD SHARING:
Plan to Share IPD: Undecided
Undecided